CLINICAL TRIAL: NCT06709144
Title: Borderline of CME/D3 Dissection for Local Advanced Right-sided Colon Cancer(BLARCC): a Prospective, Multicenter Randomized Control Clinical Trial
Brief Title: Borderline of CME/D3 Dissection for Local Advanced Right-sided Colon Cancer
Acronym: BLARCC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haixing Ju, MD (Other)
Collaborators: Jiangxi Provincial Cancer Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Liaoning Cancer Hospital & Institute (Other); The First Affiliated Hospital of Soochow University (Other); Shanxi Province Cancer Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Shaoxing People's Hospital (Other); Shaoxing Second Hospital (Other); Ningbo No. 1 Hospital (Other); Ningbo No.2 Hospital (Other); Jinhua Central Hospital (Other); Affiliated Hospital of Jiaxing University (Other); The First People's Hospital of Huzhou (Other); The Central Hospital of Lishui City (Other); Lishui Country People's Hospital (Other); Zhejiang University (Other); Yuyao People's Hospital (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Cancer Hospital of Guangxi Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Ruijin Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shanghai Cancer Hospital, China (Other); The Affiliated Tumor Hospital of Harbin Medical University (Unknown); Shanghai 10th People's Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Xiangshan No.1 People' s Hospital (Unknown); Zhejiang Province People's Hospital (Unknown); Sir Run Run Shaw Hospital (Other); Sun Yat-sen University Cancer Hosptial (Unknown)
Responsible Party: Sponsor-Investigator, Haixing Ju, MD, Director, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-935（IIT）; 2024IITZA001 (Other: Zhejiang cancer hospital)
Record Dates: First submitted 2024-11-18; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-08

CONDITIONS: Colon Cancer
Keywords: right side colon cancer; complete mesentery resection
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group SMA (Experimental): The lymph node dissection boundary is on the left side of the superior mesenteric artery (SMA).
  Interventions: Procedure: SMA lymph node dissection
- Group SMV (Active Comparator): The lymph node dissection boundary is on the left side of the superior mesenteric vein (SMV)
  Interventions: Procedure: SMV lymph node dissection

INTERVENTIONS:
Procedure: SMA lymph node dissection — The lymph node dissection boundary is on the left side of the superior mesenteric artery (SMA)
  Arms: Group SMA
Procedure: SMV lymph node dissection — The lymph node dissection boundary is on the left side of the superior mesenteric vein (SMV)
  Arms: Group SMV

SUMMARY:
The study was conducted on patients with advanced right-sided colon cancer, and the clinical pathological and prognostic data of the patients were compared between the two groups of patients who were randomly divided into those undergoing SMV and SMA left resection, with the aim of resolving the controversy over the left resection boundary of CME/D3 lymph node dissection through this study, and to clarify whether SMA left resection is superior to SMV left resection.

ELIGIBILITY:
Inclusion Criteria:

* right side colon cancer(The primary lesion is located in the ileocecal region, ascending colon, hepatic flexure of colon, or proximal transverse colon)
* T3-4 and/or N1-2M0
* Colonoscopy and pathological biopsy confirmed colon adenocarcinoma

Exclusion Criteria:

* T1-2N0M0
* Cannot undergo curative resection
* Simultaneous multiple primary colorectal cancer or other diseases requiring segmental resection
* Distant metastasis
* Tumor invades surrounding organs, requiring joint organ resection
* Emergency surgery is required for complications such as intestinal obstruction, perforation, and bleeding
* Patients who have received neoadjuvant therapy before surgery
* Pregnant or lactating women
* Patients who are not suitable or unable to tolerate surgery

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
3 year DFS | 3 years
  3 year disease free survival

SECONDARY OUTCOMES:
5 year OS | 5 years
  5 year Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Haixing Ju, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China